CLINICAL TRIAL: NCT06446050
Title: CXCL Chemokine and TNF Superfamily Co-stimulatory Molecule-modified Mesenchymal Stem Cells for the Treatment of Advanced Colorectal Cancer
Brief Title: Chemokine and Co-stimulatory Molecule-modified Mesenchymal Stem Cells for the Treatment of Advanced Colorectal Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022TILINSHEN002
Record Dates: First submitted 2024-05-29; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2023-06

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Intervention Model Description: Patients will receive infusion of MSC-L every 21 days.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC-L (Experimental): Mesenchymal Stem Cells mobilizing Lymphocytes (MSC-L)
  Interventions: Biological: MSC-L

INTERVENTIONS:
Biological: MSC-L — Human umbilical cord-derived mesenchymal stem cells (MSCs) genetically modified to express antitumor chemokine and co-stimulatory molecule will be administered intravenously at a dose of 1/2/3 x 10^6 cells/kg, every 21 days for at least 6 cycles of treatment.

SUMMARY:
The aim of this study is to assess the safety and efficacy of human umbilical cord-derived allogenic mesenchymal stem cells (MSCs) engineered to express antitumor chemokine and co-stimulatory molecule. Following systemic administration, these cells are able to migrate into solid tumors such as colorectal tumors. Once enriched in the tumor, they will attract peripheral lymphocytes consisting of T and natural killer (NK) cells, and simultaneously stimulate the infiltrated lymphocytes for persistent and enhanced antitumor immunity. Thus, this MSC-based treatment provides a potentially effective and targeted immunotherapeutic strategy for tumors with unfavorable immune microenvironment and possibly poor response to immune checkpoint blockade (ICB).

During this investigator-initiated trial (IIT), colorectal cancer patients will receive modified MSCs every 21 days via intravenous infusion. Increasing does will be tested in the initial cohort and an optimal dose will be chosen for the remaining patients.

ELIGIBILITY:
Inclusion Criteria (Participants must meet all of the following selection criteria in order to participate in this study):

1. Age less than 18 years old (including 18 years old), regardless of gender;
2. Patients with metastatic or locally advanced colorectal cancer confirmed by pathological histology or cytology;
3. According to the Efficacy Evaluation Criteria for Solid Tumors (RECIST) version 1.1, there are very few measurable tumor lesions;
4. Individuals who have progressed or are intolerant to standard treatment in the past, or patients who refuse standard treatment;
5. Severe abnormalities in the fluid system, liver and kidney function: lymphocyte count ≥ 0.8 × 10^9/L, absolute neutrophil count ≥ 1.5 × 10^9/L, hemoglobin ≥ 9g/dL, platelet count ≥ 75 × 10^9/L; Alanine aminotransferase (ALT) ≤ 3 times upper limit of normal (ULN), aspartate aminotransferase (AST) ≤ 3 times ULN, creatinine ≤ 1.5 times ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 times ULN, prothrombin time (PT) ≤ 1.5 times ULN, international standardized mean value (INR) ≤ 1.5 times ULN;
6. Eastern Cooperative Oncology Group (ECOG) score 0-2;
7. Patients with fertility must agree to use reliable contraceptive methods (hormone or barrier method or abstinence) during the trial period and at least 12 weeks after the last treatment;
8. Patients who have not undergone any other adoptive immune cell therapy or stem cell therapy within two years;
9. The patient is willing to participate and sign an informed consent form in writing.

Exclusion Criteria (Subjects with any of the following characteristics are not eligible to participate in this study):

1. Individuals with a history of allergies to biological agents or allergies to any ingredients used for cell culture;
2. Pregnant or lactating individuals;
3. Expected shelf life of more than 3 months;
4. Active infections that require systemic treatment or uncontrollable infections;
5. The adverse reactions of previous anti-tumor treatments have not yet recovered to Common Terminology Criteria for Adverse Events 4.03 (CTCAE4.03) level evaluation ≤ 1 level (excluding hair loss);
6. Have a history of severe cerebrovascular diseases, including but not limited to ventricular arrhythmias that require clinical intervention; Within 6 months, there have been acute coronary syndrome, myocardial infarction, congestive heart failure, stroke, or other Grade III or higher cardiovascular events; The New York Heart Association (NYHA) Heart Function Rating ≥ Grade II or Left Ventricular Ejection Score (LVEF) <50%; Poor control of hypertension despite standard treatment (systolic blood pressure >150mmHg, diastolic blood pressure >90mmHg);
7. A history of severe pulmonary parenchyma or pulmonary vascular related diseases, including but not limited to high-risk individuals for venous thromboembolism (VTE) (Padua score ≥ 4), as outlined in the Chinese Consensus of Cardiopulmonary Resuscitation Experts on Venous Thromboembolism Cardiac Arrest (CA) Guidelines; Or oxygen may be needed to maintain sufficient blood oxygen saturation (≥ 95%);
8. Patients with clinical symptoms of central nervous system metastasis and/or cancerous meningitis (patients with stable brain metastasis can be grouped), and those suspected of central nervous system or leptomeningeal metastasis need CT/MRI examination to rule them out;
9. Individuals with clinically confirmed autoimmune diseases (excluding thyroiditis);
10. Individuals with HIV infection; Individuals with acute Epstein-Barr virus (EBV) or cytomegalovirus (CMV) virus infection;
11. Patients with active replication of hepatitis B virus (DNA > 1000 cps/mL), hepatitis C patients;
12. Individuals who have received allogeneic bone marrow transplantation in the past;
13. Immunosuppressive subjects, including known immunodeficiencies; Within 14 days before the first dose of cell therapy and during the study period, those who require systemic use of steroid drugs (prednisone >10mg/day or equivalent doses of similar drugs) or other immunosuppressants (excluding those who have recently or recently used systemic steroids, or short-term use of steroid drugs for preventive treatment);
14. Known to have alcohol or drug dependence;
15. The researcher assessed that there may be medical history or disease, treatment or abnormal experimental values that may hinder the full participation of the subjects in this clinical study, or other situations that are not suitable for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities rate (DLT) | 4 months
  Proportion of patients who has experienced a DLT
Adverse Event (AE) | 4 months
  Proportion of patients who has experienced an AE
Determination of optimal dose of MSC-L | 4 months
  The largest dose that has an estimated risk of causing DLT (defined as MSC-L related adverse event of grade 3 or higher) equal or closest to the target level of 35% (the target toxicity level).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 24 months
  Percentage of patients cancer whose MSC-L treatment has led to a complete response, partial response, or stable disease.
Progression-free survival (PFS) | 24 months
  Time from the date of first dose of study treatment to the date of progression or death from any cause.
Overall Survival (OS) | 24 months
  Time from the date of first dose of study treatment to the date of death.
MSC-L kinetics in peripheral blood | 21 days post first infusion
  Quantification of circulating MSC-L in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Gao, MD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital (South Division), Shanghai, Shanghai Municipality, China